CLINICAL TRIAL: NCT07135180
Title: Exploring the Eye Care Benefits of Cordyceps Cicadae Across Different Age Groups
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Hui Wen Lin, Clinical Professor, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CS2-25025
Record Dates: First submitted 2025-08-11; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Visual Acuity; Accommodation; Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): Cordyceps cicadae 500mg
  Interventions: Dietary Supplement: Cordyceps cicadae
- Placebo Comparator Arm (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Blank control

INTERVENTIONS:
Dietary Supplement: Cordyceps cicadae — Cordyceps cicadae 500mg
  Arms: Experimental Arm
Dietary Supplement: Blank control — Blank control
  Arms: Placebo Comparator Arm

SUMMARY:
The aim of this study is to evaluate the underlying mechanisms of consuming two capsules (each containing 250 mg of Cordyceps cicadae mycelium, for a total intake of 500 mg) of Grape King's Cordyceps cicadae mycelium through a clinical human trial. By including participants from different age groups, the study investigates whether improvements in visual acuity and the alleviation of eye fatigue are associated with changes in ocular accommodation, tear film stability, and blood circulation. The ultimate goal is to develop a health supplement beneficial for vision.

DETAILED DESCRIPTION:
Over the past decade, vision problems caused by electronic screen use across all age groups have gradually shifted from being primarily occupational health issues to broader public health concerns. Moreover, studies have shown that prolonged computer use may lead to blurred vision at near or far distances-one of the hallmark symptoms of Computer Vision Syndrome (CVS), also known as Digital Eye Strain (DES). A key contributing factor is inaccurate accommodative response, either due to underaccommodation or overaccommodation while focusing on a visual target, leading to visual fatigue.

Sheedy et al. identified common symptoms of visual fatigue, including eye tiredness, discomfort, burning, irritation, pain, soreness, eye ache, double vision, photophobia, blurriness, itching, tearing, dryness, and a foreign body sensation. These symptoms are generally classified into two categories: the first, external symptoms-such as burning, irritation, dryness, and tearing-are associated with dry eye syndrome; the second, internal symptoms-such as eye fatigue, headache, ocular pain, diplopia, and blurred vision-are typically linked to refractive errors, accommodative dysfunction, or convergence anomalies.

In addition, a study by Tosha et al. found that subjects who experienced greater visual discomfort after prolonged computer use exhibited a significant increase in accommodative lag, suggesting a link to accommodative fatigue. Overall, these conditions are closely related to visual fatigue, and if left unmanaged, may impair visual function over time and potentially contribute to the progression of myopia.

Therefore, appropriately managing screen time, along with adequate visual rest and eye care strategies, is essential for maintaining healthy accommodation and visual function. Previous studies have demonstrated that Cordyceps cicadae mycelium can effectively relieve eye fatigue and improve visual acuity; however, the underlying mechanisms remain unclear. The Cordyceps cicadae mycelium used in this study has passed 16 safety evaluation tests and has been granted a New Dietary Ingredient (NDI No. 834) number by the U.S. Food and Drug Administration (FDA), as well as food clearance approval by Japanese customs. The product is supplied by Grape King Bio. This study aims to further investigate the eye-protective mechanisms of Cordyceps cicadae mycelium and its beneficial effects on visual health across different age groups.

ELIGIBILITY:
Inclusion Criteria:

* People with myopia less than 700 degrees
* Willing to participate in this study and sign the consent form

Exclusion Criteria:

* (1) Those who have recently consumed related eye care products
* (2) Those who have had eye infections or surgery in the past three months
* (3) Those who have been diagnosed with eye diseases by an ophthalmologist (such as glaucoma, cataracts, macular degeneration, diabetic retinopathy, etc., or have undergone eye surgery such as cataract surgery, retinal laser surgery, myopia laser surgery, etc., which will be excluded before accepting the case)
* (4) Those who are allergic to cicada fungus

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Eye fatigue questionnaire | 3 hours
  The Ocular Surface Disease Index (OSDI) was used to assess visual fatigue. The subjects were asked to fill in the questionnaire before and after taking the medicine, and the scores were calculated. Symptoms include eyestrain, discomfort, burning, irritation, pain, soreness, eye pain, double vision, photophobia, blurriness, itching, tearing, dryness, and foreign body sensation
Tear break-up time | 3 hours
  Tear film break-up time (TBUT) on the corneal surface will be recorded in seconds using corneal topography.
Accommodative Facility | 3 hours
  Use +/- 0.50D flip mirror and special optometry cards to test the number of optometry cards that the patient can read within one minute and record the number of flip cycles.
Visual acuity measurement | 3 hours
  Examinations include (a) distance visual acuity (DVA) and (b) near visual acuity (NVA), recorded using the Snellen chart.
Choroidal thickness test | 3 hours
  Heidelberg SPECTRALIS optical coherence tomography (OCT) was used to examine the choroid thickness in micrometer of the subjects.
Tear meniscus height (TMH) | 3 hours
  Tear meniscus height (TMH) will be evaluated using slit-lamp biomicroscopy and recorded in millimeters.
Meibomian gland observation | 3 hours
  The meibomian glands will be evaluated using corneal topography to document their morphology, quantity, and size.

SECONDARY OUTCOMES:
Intraocular Pressure | 3 hours
  The intraocular pressure (IOP) of the subjects was measured by non-contact intraocular pressure measurement in mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Wen Lin, Ph.D, Principal Investigator — Chung Shang medical university
Locations (1):
- Chung Shan Medical University Hui-Wen Lin lab, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No
This experiment involves patents and intellectual property rights